CLINICAL TRIAL: NCT03449173
Title: Phase II Trial of Sunitinib in Patients With Type B3 Thymoma or Thymic Carcinoma in Second and Further Lines (Style Trial)
Brief Title: Trial of Sunitinib in Patients With Type B3 Thymoma or Thymic Carcinoma in Second and Further Lines (Style Trial)
Acronym: Style
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 165-16
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Type B3 Thymoma; Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib orally administered at 50 mg once daily for 4 consecutive weeks, followed by a 2-week rest period (schedule 4/2) to comprise a complete cycle of 6 weeks
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — small-molecule, multi-targeted receptor tyrosine kinase (RTK) inhibitor
  Other Names: Sutent

SUMMARY:
Study to investigate response to sunitinib in patients with thymic epithelial tumours who had progressive disease after at least one previous regimen of platinum-based chemotherapy.

DETAILED DESCRIPTION:
This trial will be conducted to assess the activity of Sunitinib in patients affected by advanced or recurrent B3 thymoma or thymic carcinoma progressing after at least one line of chemotherapy (including one platinum based regimen).

Taking into account the different biology and historically discrepant responses and survival of thymoma and thymic carcinoma, patients will be enrolled with these tumour types in two separate cohorts.

Sunitinib will be self orally administered at 50 mg once daily, is 50 mg taken orally once daily, for 4 consecutive weeks, followed by a 2-week rest period (schedule 4/2) to comprise a complete cycle of 6 weeks until tumour progression, unacceptable toxicity or other criteria for discontinuation is met.

Sunitinib dose reductions are permitted as per the approved product label for safety reasons.

Dose reductions should occur in 12.5 mg decrements. No more than 2 dose reductions are allowed. If more than 2 dose reductions are necessary (ie, reduction to less than 25 mg daily), the subject must be permanently discontinued (Section 7.2.2)

Possible dose reductions:

* Sunitinib at dose of 37,5 mg orally once daily for 4 weeks followed by 2 weeks rest-period in cycles of 6 weeks.
* Sunitinib at dose of 25 mg orally once daily for 4 weeks followed by 2 weeks rest-period in cycles of 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IRB (Independent Review Board)/IEC (Independent Ethics Committee)-approved Informed Consent
2. Histological diagnosis of invasive recurrent or metastatic type B3 thymoma or thymic carcinoma. In case of presence of both histologies it will be classified based on the predominantly part. B2 thymoma with areas of B3 thymoma are eligible.
3. Patients must have had at least one prior platinum-containing chemotherapy regimen. There is no limit to the number of prior chemotherapy regimens or targeted agents received. Progressive disease should have been documented before entry into the study
4. Patients must have measurable disease, defined as at least one lesion that can be accurately measured according with RECIST 1.1 criteria
5. Availability of archival tissue (paraffine block or at least 10 unstained slides)
6. Patients must have recovered from toxicity related to prior therapy to at least grade 1 (defined by v.CTCAE 4.0)
7. Patients must not have had major surgery, radiation therapy, chemotherapy, biologic therapy (including any investigational agents), or hormonal therapy (other than replacement), within 4 weeks prior to entering the study
8. Age > 18 years
9. Life expectancy > 3 months
10. Performance status (ECOG) ≤ 2
11. Negative pregnancy test (if female in reproductive years)
12. Patients must have adequate organ and marrow function (as defined below). Patients must have returned to baseline or grade 1 from any acute toxicity related to prior therapy:

    * Absolute neutrophil count ≥ 1,500/mm
    * Hemoglobin ≥ 9 g/dL
    * Platelets ≥ 100,000/mm
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) , except for patients affected by Gilbert's syndrome
    * AST(SGOT) (aspartate aminotransferase) /ALT(SGPT) (alanine transaminase) ≤ 3 x institutional ULN (5x if LFT (liver function test) elevations due to liver metastases)
    * Creatinine ≤ 1.5 x institutional ULN
13. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception before study entry, for all the duration of the study and for at least 8 weeks after the last dose of investigational drug (30 days for an ovarian cycle turnover plus the time required for the active metabolite of sunitinib to undergo five half-lives).
14. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of before study entry, for all the duration of the study and for at least 16 weeks after the last dose of investigational drug (90 days for sperm turnover plus the time required for the active metabolite of sunitinib to undergo five half-lives).

Exclusion Criteria:

1. untreated CNS metastases. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to start of treatment, or after surgical resection performed at least 28 days prior to start of treatment. The patient may have no evidence of Grade ≥1 CNS haemorrhage based on pre-treatment Magnetic Resonance Imaging (MRI) or IV contrast CT scan (performed within 28 days before start of treatment)
2. Major surgery, other than diagnostic surgery, within 4 weeks prior to treatment
3. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
4. Pregnant or breast feeding women
5. Previous (within the last 5 years) or current malignancies at other sites, except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri
6. Current enrollment in or participation in another therapeutic clinical trial within 4 weeks before treatment start.
7. Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months, unstable angina within 6 months, NYHA (New York Heart Association) Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%,
8. Ongoing symptomatic cardiac dysrhythmias, uncontrolled atrial fibrillation, or prolongation of the Fridericia corrected QT (QTcF) interval defined as > 450 msec for males and > 470 msec for females, where QTcF = QT / 3√RR
9. Poorly controlled hypertension
10. History of cerebrovascular accident including transient ischemic attack within the past 12 months.
11. History of deep vein thrombosis (DVT) unless adequately treated with low molecular weight heparin
12. History of pulmonary embolism within the past 6 months unless stable, asymptomatic, and treated with low molecular weight heparin for at least 6 weeks.
13. Evidence of active bleeding or bleeding susceptibility; or medically significant hemorrhage within prior 30 days.
14. Receiving concomitant CYP3A4 inducers or strong CYP3A4 inhibitors
15. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sunitinib
16. Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Activity of Sunitinib | 4 years
  Best tumour response (Complete Response + Partial Response)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 4 years
  The PFS is defined as the time from the date of randomization to the date of documented progressive disease, recurrence or Death (whichever occurs first)
Overall Survival (OS) | 4 years
  The OS is defined as the time from the date of randomization to the date of death
Duration of activity of sunitinib | 4 years
  Complete Response + Partial Response + Stable Disease
Safety and toxicity profile of sunitinib | 4 years
  will be utilized the CTCAE v 4.0 criteria for assessment of toxicity and serious adverse event reporting.
Incidence of adverse events (AEs) | 4 years
  Incidence of adverse events (AEs) will be graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0, laboratory values, physical examinations, vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Chiara Garassino, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurup A et al. Phase II study of gefitinib treatment in advanced thymic malignancies. JCO 23 (16S, Part I of II, June 1 Supplement), ASCO 2005: Abs. 7068
- [Background] Thomas A, Rajan A, Berman A, Tomita Y, Brzezniak C, Lee MJ, Lee S, Ling A, Spittler AJ, Carter CA, Guha U, Wang Y, Szabo E, Meltzer P, Steinberg SM, Trepel JB, Loehrer PJ, Giaccone G. Sunitinib in patients with chemotherapy-refractory thymoma and thymic carcinoma: an open-label phase 2 trial. Lancet Oncol. 2015 Feb;16(2):177-86. doi: 10.1016/S1470-2045(14)71181-7. Epub 2015 Jan 13. PMID 25592632
- [Background] Salter JT et al. Imatinib for the treatment of thymic carcinoma. JCO 26: ASCO 2008 (May 20 Supplement): Abs.
- [Result] Engels EA, Pfeiffer RM. Malignant thymoma in the United States: demographic patterns in incidence and associations with subsequent malignancies. Int J Cancer. 2003 Jul 1;105(4):546-51. doi: 10.1002/ijc.11099. PMID 12712448
- [Result] Wright CD. Management of thymomas. Crit Rev Oncol Hematol. 2008 Feb;65(2):109-20. doi: 10.1016/j.critrevonc.2007.04.005. Epub 2007 Jun 14. PMID 17570676
- [Result] Giaccone G. Treatment of malignant thymoma. Curr Opin Oncol. 2005 Mar;17(2):140-6. doi: 10.1097/01.cco.0000152628.43867.8e. PMID 15725919
- [Result] Serpico D, Trama A, Haspinger ER, Agustoni F, Botta L, Berardi R, Palmieri G, Zucali P, Gallucci R, Broggini M, Gatta G, Pastorino U, Pelosi G, de Braud F, Garassino MC. Available evidence and new biological perspectives on medical treatment of advanced thymic epithelial tumors. Ann Oncol. 2015 May;26(5):838-847. doi: 10.1093/annonc/mdu527. Epub 2014 Nov 19. PMID 25411417
- [Result] Strobel P, Hartmann M, Jakob A, Mikesch K, Brink I, Dirnhofer S, Marx A. Thymic carcinoma with overexpression of mutated KIT and the response to imatinib. N Engl J Med. 2004 Jun 17;350(25):2625-6. doi: 10.1056/NEJM200406173502523. No abstract available. PMID 15201427
- [Result] Bisagni G, Rossi G, Cavazza A, Sartori G, Gardini G, Boni C. Long lasting response to the multikinase inhibitor bay 43-9006 (Sorafenib) in a heavily pretreated metastatic thymic carcinoma. J Thorac Oncol. 2009 Jun;4(6):773-5. doi: 10.1097/JTO.0b013e3181a52e25. PMID 19461405